CLINICAL TRIAL: NCT03393702
Title: Efficacy of Gabapentin as Adjuvant for Postoperative Pain in Pediatric Thoracic Surgery - a Randomized Quadruple Blind Study
Brief Title: Pain Control in Children and Adolescent After Thoracic Surgery: The Effect of Gabapentin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute for Tuberculosis and Lung Diseases, Poland (Other)
Responsible Party: Principal Investigator, Lucyna Tomaszek, PhD, RN, Head of Nursing, Specialist Nurse in Anesthesia and Intensive Care, National Institute for Tuberculosis and Lung Diseases, Poland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10.11
Record Dates: First submitted 2017-12-28; First posted 2018-01-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Pain, Postoperative; Surgery, Thoracic
Keywords: Postoperative pain; Anxiety; Postoperative Complications; Patient Satisfaction
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Postoperative Complications; Patient Satisfaction | interventions — Gabapentin; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Experimental): 1. Single dose preoperative gabapentin.
  2. After surgery gabapentin 2 times per day for 3 days.
  Interventions: Drug: Gabapentin
- Placebo Control (Placebo Comparator): 1. Single dose preoperative placebo control.
  2. After surgery placebo 2 times per day for 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — 1. Patients in this arm of the study receive identical capsules, containing 15 mg/kg of oral gabapentin.
  2. Patients after surgery receive identical capsules, containing 7,5 mg/kg of oral gabapentin 2 times per day.
  Other Names: Gabapentin TEVA, capsules
  Arms: Gabapentin
Drug: Placebo — 1. Patients in this arm of the study receive identical placebo capsules 1 hour before surgery.
  2. Patients after surgery receive identical placebo capsules 2 times per day.
  Arms: Placebo Control

SUMMARY:
The study is performed in patients aged 5-18 years after thoracic surgery. The primary aim of this trial is to determine whether the use of gabapentin as a component of multimodal analgesic regiments reduces pain scores following thoracic surgery in pediatric patients. The secondary objective of the trial are to evaluate whether the use of gabapentin reduces postoperative anxiety scores and consumption of ropivacaine with fentanyl, decreases side-effects, and improves patient satisfaction.

DETAILED DESCRIPTION:
The subjects are randomized to the Gabapentin or Placebo group. All patients receive preoperative gabapentin (15 mg/kg, treatment) or placebo, respectively and after surgery either gabapentin (7,5 mg/kg, treatment) or placebo 2 times per day for 3 days, respectively.

Patients are subjected to the same anaesthesia protocol. Postoperative analgesia are achieved with either continuous ropivacaine 0.2%/fentanyl 5.0 μg/ml infusion through a thoracic epidural catheter (N=40; Gabapentin n=20, Placebo n=20), or intravenous infusion of morphine (N=40; Gabapentin n=20, Placebo n=20). All patients receive acetaminophen and non-steroidal anti-inflammatory drugs, and metamizol as a "rescue drug"

The intravenous infusion of morphine grup was expanded on the basis of the bioethics commission's decision KB-125/2019 (N=64; Gabapentin n=32, Placebo n=32).

ELIGIBILITY:
Inclusion Criteria:

* 5 - 18 years of age;
* surgery: lateral thoracotomy or Ravitch procedure;
* ASA 1-3;
* postoperative analgesia: thoracic epidural analgesia or intravenous infusion of morphine.

Exclusion Criteria:

* allergy or sensitivity to gabapentin;
* history of chronic pain or daily analgesic use;
* diagnosed with psychiatric disorders;
* treated oncologically;
* with impaired verbal communication;
* the lack of postoperative chest drainage.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity scores at rest (FLACC for patients <7 y.o., NRS for patients >7 y.o.) | postoperative day: 0-3
Pain intensity scores during deep breathing (FLACC for patients <7 y.o., NRS for patients >7 y.o.) | postoperative day: 0-3
Pain intensity scores during coughing (FLACC for patients <7 y.o., NRS for patients >7 y.o.) | postoperative day: 0-3

SECONDARY OUTCOMES:
Total ropivacaine/fentanyl consumption. | postoperative day: 0-3
Total morphine consumption. | postoperative day: 0-3
Anxiety intensity scores. | before surgery, postoperative day 3
  Patients rate their anxiety using State-Trait Anxiety Inventory.
Side Effect Occurrence | first 3 days after surgery
  Incidence and severity of nausea, vomiting, pruritis, sedation, dizziness, urinary retention, complication in relation to administering of the drugs to epidural space.
The number of doses of metamizol as a "rescue drug" | postoperative day: 0-3
Patient satisfaction. | first 3 days after surgery
  Responses can range from 0 (very dissatisfied) to 10 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Lucyna Tomaszek, PhD, Study Director — National Institute for Tuberculosis and Lung Diseases, Poland
Locations (1):
- Institute for Tuberculosis and Lung Diseases, Pediatric Division, Rabka-Zdrój, Małopolska, Poland

REFERENCES:
- [Background] Rusy LM, Hainsworth KR, Nelson TJ, Czarnecki ML, Tassone JC, Thometz JG, Lyon RM, Berens RJ, Weisman SJ. Gabapentin use in pediatric spinal fusion patients: a randomized, double-blind, controlled trial. Anesth Analg. 2010 May 1;110(5):1393-8. doi: 10.1213/ANE.0b013e3181d41dc2. PMID 20418301
- [Background] Mayell A, Srinivasan I, Campbell F, Peliowski A. Analgesic effects of gabapentin after scoliosis surgery in children: a randomized controlled trial. Paediatr Anaesth. 2014 Dec;24(12):1239-44. doi: 10.1111/pan.12524. Epub 2014 Sep 17. PMID 25230144
- [Background] Tomaszek L, Fenikowski D, Maciejewski P, Komotajtys H, Gawron D. Perioperative Gabapentin in Pediatric Thoracic Surgery Patients-Randomized, Placebo-Controlled, Phase 4 Trial. Pain Med. 2020 Aug 1;21(8):1562-1571. doi: 10.1093/pm/pnz207. PMID 31596461
- [Derived] Fenikowski D, Tomaszek L. Factors Related to Anxiety in Paediatric Patients and Their Parents before and after a Modified Ravitch Procedure-A Single-Centre Cohort Study. Int J Environ Res Public Health. 2022 Dec 12;19(24):16701. doi: 10.3390/ijerph192416701. PMID 36554581